CLINICAL TRIAL: NCT05546190
Title: Non-interventional Study to Assess the Arm Activity Measure Questionnaire (ArmA) by Patients With Adult Upper Limb (AUL) Spasticity.
Brief Title: A Study to Collect Participants Experience of Living With Adult Upper Limb (AUL) Spasticity and to Assess the Arm Activity Measure (ArmA)
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-10200-450
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Spastic Hemiparesis; Muscle Spasticity
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The participants of this study will have AUL spasticity and have a need for botulinum toxin type A injections. AUL spasticity is where people develop tightening or stiffness of the muscles in the arms. Botulinum toxin type A is used for the treatment of spasticity in addition to physiotherapy. This study will ask participants to describe their experience living with AUL spasticity. This information will be used to assess the Arm Activity Measure (ArmA). ArmA is a scale designed to assess upper limb function in people with AUL spasticity. This study could suggest changes to the ArmA to improve its suitability for people with AUL spasticity or even the development of a new scale.

ELIGIBILITY:
Inclusion Criteria :

* Participant has provided informed consent and is willing to take part in the study
* Participant is an adult aged at least 18 years
* Participant has a clinical diagnosis of spastic hemiparesis following stroke or traumatic brain injury (TBI) affecting one arm only
* Participant is at least 6 months post-stroke or TBI
* Participant has a need for botulinum toxin type A injections as part of their treatment for AUL spasticity
* Patient is considered to be in a stable state with regard to their therapeutic interventions (i.e., all treatments for the patient's condition have been stable for at least one month prior to assessment of eligibility)
* Participant has access to the internet, laptop, or tablet, and is willing to take part in either an online focus group or interview (caregiver assistance is acceptable)
* Participant is fluent in the English language and is able to discuss their condition

Exclusion Criteria :

* Participant has any medical condition that prohibits their ability to communicate with the interviewer including severe dysphasia or an inability to read questionnaires.
* Participant has any other clinically relevant concern (e.g., significant psychiatric disorder or depression, history of alcohol and/or drug abuse) that in your opinion would interfere with their ability to provide written informed consent and/or participate.
* Participant has AUL spasticity is present in both arms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are at least 18 years old, able to read and communicate fluently in English and have a clinical diagnosis of spastic hemiparesis following stroke or traumatic brain injury (TBI). They must be at least 6 months post-stroke or TBI and have AUL in both arms that requires botulinum toxin type A injections as part of their AUL spasticity treatment.
  Additionally, participants are required to be in a stable state regarding their therapeutic interventions (i.e., at least one month prior to assessment of eligibility) and have no other clinically relevant concerns that would hinder their ability to provide written informed consent and/or participate.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Number of participants answering to the questionnaire: for Part 1 15/15 subject | First interview/ at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (2):
- United States (2):
  - Rancho Los Amigos National Rehab, Downey, California
  - MedStar National Rehabilitation Network, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/